CLINICAL TRIAL: NCT05712473
Title: A Prospective Observational Multicenter Real-World Registry Assessing the Impact of the Use of PYLARIFY® (Piflufolastat F18) PET in Patients With Prostate Cancer
Brief Title: An Observational Registry Assessing the Impact of PYLARIFY® (Piflufolastat F18) PET in Patients With Prostate Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Specialty Networks Research. (Network)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-403
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients who are newly diagnosed with prostate cancer (and have suspected metastases) and have not yet initiated any prostate cancer treatment and are referred to undergo PYLARIFY PET
  Interventions: Diagnostic Test: PYLARIFY
- Cohort 2:: Patients who have previously received treatment for prostate cancer and are referred to undergo PYLARIFY PET or have received PYLARIFY PET for suspected recurrence of prostate cancer (based on an elevated PSA) within 60 days of consent to enroll in the registry
  Interventions: Diagnostic Test: PYLARIFY

INTERVENTIONS:
Diagnostic Test: PYLARIFY — PYLARIFY PET

SUMMARY:
The goal of this observational research is to assess the real-world clinical utility of PYLARIFY PET through evaluation of long-term outcomes for prostate cancer patients who are eligible for a PSMA/PET scan.

Participants will be enrolled at their physician's office at the time of referral for PYLARIFY PET and will be followed for up to 5 years. Data concerning their prostate cancer diagnostics and treatment will be collected at 6-month intervals.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following inclusion criteria:

1. Biological male at birth ≥ 21 years of age
2. Histopathological confirmed prostate adenocarcinoma
3. Patients meeting the enrollment criteria for either Cohort 1 or Cohort 2:

   1. Cohort 1:

      Patients who are newly diagnosed with prostate cancer (and have suspected metastases per the physician's discretion per standard of care assessment) and have not yet initiated any prostate cancer treatment and are referred to undergo PYLARIFY PET for identification of suspected metastases.

      OR
   2. Cohort 2:

   Patients who have previously received treatment for prostate cancer and are referred to undergo PYLARIFY PET or have received PYLARIFY PET for suspected recurrence of prostate cancer (based on an elevated PSA) within 60 days of consent to enroll in the registry
4. Life expectancy ≥ 6 months as determined by the investigator
5. Able and willing to provide informed consent and comply with the protocol requirements.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not eligible for enrollment in this study:

1. Patients who are referred for PSMA PET and undergo a PSMA PET with a radioactive agent other than PYLARIFY
2. Patients who have histological evidence of neuroendocrine prostate cancer (NEPC) (small cell/ductal variant)
3. Patients with any medical condition or other circumstances that, in the opinion of the investigator, compromise the safety of compliance of the patient to produce reliable data or completing the study.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Registry is specifically for prostate cancer patients (limited to biologically male).
Study Population: Biologically male patients with confirmed prostate cancer referred to undergo a PSMA PET with PYLARIFY.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 5 years
  The objective of this registry is to assess the real-world clinical utility of PYLARIFY PET through evaluation of long-term outcomes for prostate cancer patients who are eligible for a PSMA/PET scan and for whom PYLARIFY imaging is incorporated into treatment recommendations and management plans.

SECONDARY OUTCOMES:
Secondary Objective 1 | 5 years
  To understand the demographic and clinical characteristics of patients referred for PYLARIFY PET.
Secondary Objective 2 | 5 years
  To understand the impact of PYLARIFY PET results on healthcare resource utilization.
Secondary Objective 3 | 5 years
  To understand the role of PYLARIFY PET in treatment change management for newly diagnosed prostate cancer patients.
Secondary Objective 4 | 5 years
  To understand the utilization of PYLARIFY PET at very low PSA levels in patients with oligometastatic prostate cancer.
Secondary Objective 5 | 5 years
  To understand racial and ethnic disparities in prostate cancer care.